CLINICAL TRIAL: NCT01409889
Title: Comparative Effectiveness of Practice-Based Diabetes Prevention Programs - A Pilot Study
Brief Title: Comparing Diabetes Prevention Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Nancy Bennett, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CTSI 5-27805
Record Dates: First submitted 2011-08-02; First posted 2011-08-04 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Pre Diabetes; Diabetes
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diabetes Prevetion Program (Active Comparator): Individuals in this group will receive the Diabetes Prevention Program
  Interventions: Behavioral: Diabetes Prevention Program
- Healthy Living Program (Active Comparator): Individuals in this group will receive the Healthy Living Program
  Interventions: Behavioral: Healthy Living Program

INTERVENTIONS:
Behavioral: Diabetes Prevention Program
  Other Names: DPP
  Arms: Diabetes Prevetion Program
Behavioral: Healthy Living Program
  Other Names: HLP
  Arms: Healthy Living Program

SUMMARY:
The purpose of this study is to compare the effectiveness and costs of two programs,the Diabetes Prevention Program and the community-developed Healthy Living Program, delivered in an primary care practice.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* diagnosed with pre-diabetes

Exclusion Criteria:

* diagnosed with diabetes
* pregnant or nursing
* unable to walk 2-3 blocks in 10 minutes
* unable to read and speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2011-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Participant Weight | 22 weeks
  7% reduction in participant weight

SECONDARY OUTCOMES:
Minutes of Physical Activity | 22 weeks
  Increase physical activity to 150 minutes per week.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Anthony Jordan Health Center, Rochester, New York
  - Rochester General Medical Associates, Rochester, New York
  - Unity Health System, Rochester, New York
  - Westside Health Services, Rochester, New York